CLINICAL TRIAL: NCT03858816
Title: Efficacy of Multiple Strain Probiotics Reduces the Neurobehavioral Disorder in Premature Very Low Birth Weight Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting participants.
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hung-Chih Lin, Attending physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH106-REC2-102
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Very Low Birth Weight Infants
Keywords: probiotics; neuropsychiatric disorder; very low birth weight infants; attention deficit and hyperactivity disorder (ADHD); autism spectrum disorder (ASD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixture probiotics (Experimental): The probiotic contain 1 ×10^9 CFU/1 capsule of mixture probiotics, taking 1 probiotic capsule for up to 4 months after birth.
  Interventions: Other: Mixture probiotics
- Placebo (Placebo Comparator): Taking 1 placebo capsule for up to 4 months after birth.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Mixture probiotics — The mixture probiotics capsule
  Arms: Mixture probiotics
Other: Placebo — The placebo contains the same excipient ingredients but without the live bacteria.
  Arms: Placebo

SUMMARY:
The management protocols, clinical practices, equipment, infrastructure, and key personnel in NICU are unchanged during the study period. The data collected by each center are transmitted to the office of the principal investigator (Dr Lin) at China Medical University Hospital. Primary outcome is death or attention deficit and hyperactivity disorder (ADHD) and ASD.

DETAILED DESCRIPTION:
Over the years, preterm very low birth weight (PVLBW) infants (<32 weeks gestation) have better survival rates and improved outcomes. Nonetheless, It is of concern that there are increased risk of psychiatric problems reported in PVLBW infants, 11.5% to 31% of them are reported to be at increased risk of attention deficit and hyperactivity disorder (ADHD) and 25 % of them would develop autism spectrum disorder (ASD).

Many VLBWs experience rapid vaginal or Caesarean births that increased relative risk of developing ASD and possibly ADHD when compared to vaginal delivery. Further, PVLBW infants often experience delays in enteral feeding, and many receive little or no mother's own milk, use of antibiotics, invasive procedures and maternal separation can contribute to dysbiosis and dysbiosis in early life may prone to develop ASD and ADHD There is growing body of evidence demonstrates that gut microbiota is involved in communication, and may impact brain development and modulate behavior. Evidences have showed that there were increased intestinal permeability, altered gut microbiota and activity in autism and ADHD. Studies have demonstrated that early postnatal phase of microbial development is a primer for future health. Giving all the evidence, it is reasonable to speculate that probiotics could reduce the ASD and ADHD in preterm VLBW infants.

From Aug 1, 2017 to June 30, 2020, a prospective, double blind, randomized, controlled trial will be conducted in five NICUs at Taiwan. The study protocol will be approved by the institutional review board of each hospital. Preterm infants ≧ 23 weeks and ≦ 32 weeks gestational age and birth weight below 1500 gm and who survive to NICU are eligible for the trial. They will be assigned randomly to either group A: multiple strian probiotics or group B: control group received 1 mL of a 5% glucose solution. Study is continuous until preterm infants grow up to 4 months postnatal age.

The management protocols, clinical practices, equipment, infrastructure, and key personnel in NICU are unchanged during the study period. The data collected by each center are transmitted to the office of the principal investigator (Dr Lin) at China Medical University Hospital. Primary outcome is death or attention deficit and hyperactivity disorder (ADHD) and ASD.

Mortality is defined as death prior to discharge. Secondary outcomes are NEC ≧ stage 2, sepsis, severe (grade 3-4) IVH, BPD, alteration of liver function, and adverse effects or intolerance and neurodevelopment impairment. Objection of the first two years is to enroll cases, ASD and ADHD will be assessed by two independent neurologists at third year of life; no examiner is aware of treatment assigned to any infant.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants ≧ 23 weeks and ≦ 32 weeks gestational age.
* Birth weight below 1500 gm and who survive to NICU.

Exclusion Criteria:

* Severe asphyxia (stage III)
* Fetal chromosomal anomalies
* Cyanotic congenital heart disease
* Congenital intestinal atresia
* Gastroschisis
* Omphalocele
* Active upper gastric intestinal bleeding
* Lacking/refused of parental consent
* Early onset sepsis (before the third day of life)
* Liver failure (aspartate aminotransferase, alanine aminotransferase, glutamyl transferase, direct bilirubin serum values 3-fold higher than reference range)
* Fasted for >3 weeks.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of death or ADHD and ASD | Two years

SECONDARY OUTCOMES:
Incidence rate of NEC ≧ stage 2, sepsis, severe (grade 3-4) IVH, BPD, liver function and adverse effects or intolerance and neurodevelopment impairment. | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Children Hospital, China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- See also: Related Info — http://www.cmuh.cmu.edu.tw/